CLINICAL TRIAL: NCT00935337
Title: A Pilot Study of Two Contrasting Intervention Programs for Sleep Management - Part II
Brief Title: Follow-up of a Study Examining Sleep Management in United States Veterans
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Gavin West, M.D., VA Medical Center/University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 34556
Record Dates: First submitted 2009-06-18; First posted 2009-07-09 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-11

CONDITIONS: Insomnia
Keywords: Sleep problems; Awareness training program; Mind body bridging
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Parasomnias

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mind-Body Bridging Program (Experimental): Mind Body Bridging subjects will be accessed with questionnaires and medical history evaluations for the impact of MBBP over the past 6 months since undertaking the program.
  Interventions: Behavioral: Mind-Body Bridging Program
- Sleep Hygiene (Active Comparator): Sleep Hygiene subjects will be accessed with questionnaires and medical history evaluations for the impact of SH over the past 6 months since undertaking the program.
  Interventions: Behavioral: Sleep Hygiene

INTERVENTIONS:
Behavioral: Mind-Body Bridging Program — Bridging aims to reduce the impact of negative thought patterns that contribute to stress in the body.
  Other Names: MBBP
  Arms: Mind-Body Bridging Program
Behavioral: Sleep Hygiene — treatment as usual
  Other Names: SH
  Arms: Sleep Hygiene

SUMMARY:
The first part of the pilot study, as detailed in Unique Protocol ID No. 27522, is a randomized clinical trial that compares the effects of a mind-body bridging program with a sleep hygiene program to improve sleep quality in patients suffering from sleep disturbances. In Part II of the study, the investigators will perform a six month follow-up on the same subjects.

DETAILED DESCRIPTION:
In this follow-up, we ask subjects to answer the same questionnaires that they completed at the beginning of the study. In addition we will ask subjects to complete a survey reflecting their medical history over the past 6 months and a second survey establishing their behavioral patterns and whether they continued practicing techniques of the intervention they were assigned to.

ELIGIBILITY:
Inclusion Criteria:

* Have participated in Part I of this study

Exclusion Criteria:

* The patient presents with significant mental health issues, such as severe psychosis or major depression (as verified by the primary care provider) or the patient is under intensive mental health case management.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-04; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Medical Outcomes Study-Sleep Scale | 6 months following study part I
Medical Outcomes Study Short Form-36 | 6 months following study part I

SECONDARY OUTCOMES:
Center for Epidemiologic Studies Depression Scale | 6 months following study part I
Five-factor Mindfulness Questionnaire | 6 months following study part I
PTSD Check List-Military | 6 months following study part I

CONTACTS AND LOCATIONS:
Overall Officials: Gavin West, M.D., Principal Investigator — Salt Lake City VA/University of Utah
Locations (1):
- SLC VA Medical Center, Salt Lake City, Utah, United States